CLINICAL TRIAL: NCT03816475
Title: Hypofractionated 5x5 Gy Radiotherapy With Prolonged Gap Before Surgery in Preoperative Treatment of Patients With Locally Advanced Myxoid Liposarcomas of Extremities or Trunk Wall
Brief Title: Hypofractionated Radiotherapy in Locally Advanced Myxoid Liposarcomas of Extremities or Trunk Wall (LIPO-MYX Trial)
Acronym: LIPOMYX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIPOMYX1
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-01

CONDITIONS: Myxoid Liposarcoma
Keywords: Dose Hypofractionation; Neoadjuvant Therapy; Sarcoma; Dose Fractionation; Dose-Response Relationship
MeSH Terms: conditions — Liposarcoma, Myxoid; Sarcoma | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated radiotherapy (Experimental): 5x5 Gy radiotherapy and delayed surgery (after 6-8 weeks)
  Interventions: Radiation: Hypofractionated radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — Preoperative hypofractionated 5x5 Gy radiotherapy (5 consecutive days) prescribed on planned target volume (tumor volume + elective margins + setup/error margin) with daily image guidance.
  Other Names: 5x5 Gy

SUMMARY:
After a screening, which consists of pathology confirmation, physical examination, magnetic resonance imaging (MRI), body computed tomography (CT) scan, blood tests, and case analysis on Multidisciplinary Team (MDT) meeting, patient will be irradiated 5x5 Gy and after radiotherapy and then referred for surgery 6-8 weeks after the radiotherapy completion.

DETAILED DESCRIPTION:
Myxoid liposarcoma has been reported to be more radiosensitive compared with other soft tissue sarcomas (STS). Response to preoperative treatment involves in decrease in tumor size, a large percentage in tumor necrosis (which according to some reports has a beneficial effect on the reduction of local recurrence rates) and also among other in a change in vasculature of the tissue.

Hypofractionation represents a variation of radiotherapy fractionation in which the total dose is divided into fewer fractions with an increased fraction dose. Such treatment may lead to additional biological effects when compared to conventionally fractionated radiotherapy (eg. vascular damage, increased immunogenicity, and antigenicity). The main advantages of hypofractionation are those related to the decreased overall treatment time what is more convenient for both patients and physicians, increased compliance and makes the treatment more cost-effective. Intriguing, such an approach may provide an additional benefit when treating non-radiosensitive tumors with a low alpha/beta ratio (eg. sarcomas).

The use of preoperative hypofractionated radiotherapy 5x5 Gy for five consecutive days, and then immediate surgery in patients with locally advanced soft tissue sarcomas showed in a published study a good local control rate, with a favorable amount of late toxicities. In this patient population, there were 22 patients with primary myxoid liposarcoma and the local control rate in this group was 86%.

In the proposed study we plan to increase the gap between the end of radiotherapy and surgery to commonly applied five weeks to better assess the changes occurring in the tumor after treatment and to evaluate the impact of longer treatment interval on reducing the proportion of early complications of treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old;
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2;
* pathologically confirmed diagnosis of localized, potentially resectable myxoid liposarcoma;
* primary tumor without previous treatment;
* extremity or trunk wall localization of the tumor;
* eligibility for limb-sparing surgery;
* >= 5cm in the longest diameter at imaging staging (MRI);
* adequate hematologic, liver, and renal function;
* women of childbearing potential must have a negative pregnancy test on the day of registration for study;
* female subjects who are breastfeeding should discontinue nursing prior to the first day of study treatment and during the whole radiotherapy treatment;
* no co-existing malignancy within the last 2 years except for adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix;
* the absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before randomization in the trial;
* before patient randomization, written informed consent must be given according to ICH/GCP.

Exclusion Criteria:

* history of radiation to the affected volume;
* previous or planned neoadjuvant chemotherapy;
* contraindications to radiotherapy, or surgery;
* metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2015-04-24 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Wound complication rate | 6 months
  Wound complication rate

SECONDARY OUTCOMES:
Percentage of tumor necrosis | 2 months
Local control rate | 60 months
  Local control rate at 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Sklodowska-Curie Institute - Oncology Center, Warsaw, Mazovian, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kosela-Paterczyk H, Szacht M, Morysinski T, Lugowska I, Dziewirski W, Falkowski S, Zdzienicki M, Pienkowski A, Szamotulska K, Switaj T, Rutkowski P. Preoperative hypofractionated radiotherapy in the treatment of localized soft tissue sarcomas. Eur J Surg Oncol. 2014 Dec;40(12):1641-7. doi: 10.1016/j.ejso.2014.05.016. Epub 2014 Sep 20. PMID 25282099
- [Background] Chung PW, Deheshi BM, Ferguson PC, Wunder JS, Griffin AM, Catton CN, Bell RS, White LM, Kandel RA, O'Sullivan B. Radiosensitivity translates into excellent local control in extremity myxoid liposarcoma: a comparison with other soft tissue sarcomas. Cancer. 2009 Jul 15;115(14):3254-61. doi: 10.1002/cncr.24375. PMID 19472403
- [Background] Messiou C, Bonvalot S, Gronchi A, Vanel D, Meyer M, Robinson P, Morosi C, Bloem JL, Terrier PH, Lazar A, Le Pechoux C, Wardelman E, Winfield JM, Boulet B, Bovee J, Haas RL. Evaluation of response after pre-operative radiotherapy in soft tissue sarcomas; the European Organisation for Research and Treatment of Cancer-Soft Tissue and Bone Sarcoma Group (EORTC-STBSG) and Imaging Group recommendations for radiological examination and reporting with an emphasis on magnetic resonance imaging. Eur J Cancer. 2016 Mar;56:37-44. doi: 10.1016/j.ejca.2015.12.008. Epub 2016 Jan 20. PMID 26802529
- [Background] Kosela-Paterczyk H, Szumera-Cieckiewicz A, Szacht M, Haas R, Morysinski T, Dziewirski W, Prochorec-Sobieszek M, Rutkowski P. Efficacy of neoadjuvant hypofractionated radiotherapy in patients with locally advanced myxoid liposarcoma. Eur J Surg Oncol. 2016 Jun;42(6):891-8. doi: 10.1016/j.ejso.2016.02.258. Epub 2016 Mar 18. PMID 27026512